CLINICAL TRIAL: NCT03448016
Title: Linking Nociceptive Opioid Peptide (NOP) Receptors With Relapse in Alcoholism
Brief Title: [C-11]NOP-1A and Alcohol Use Disorder
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Rajesh Narendran (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor-Investigator, Rajesh Narendran, Visiting Professor in Radiology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PRO16030103 & PRO13080387; R01AA025247 (NIH)
Record Dates: First submitted 2018-02-21; First posted 2018-02-27 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — 3-alpha-Hydroxysteroid Dehydrogenase (B-Specific); 3-(2'-fluoro-6',7'-dihydrospiro(piperidine-4,4'-thieno(3,2-c)pyran)-1-yl)-2-(2-fluorobenzyl)-N-methylpropanamide

STUDY DESIGN:
Intervention Model Description: [C-11]NOP-1A
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Alcohol use disorders (Experimental): [C-11]NOP-1A PET Scan
  Interventions: Radiation: [C-11]; Drug: NOP-1A
- Controls (Experimental): [C-11]NOP-1A PET Scan
  Interventions: Radiation: [C-11]; Drug: NOP-1A

INTERVENTIONS:
Radiation: [C-11] — Radiolabel
Drug: NOP-1A — Tracer

SUMMARY:
The goal of this study is to compare [C-11]NOP-1A binding in recently abstinent alcohol use disorders and controls

DETAILED DESCRIPTION:
This will allow for understanding brain stress and antistress mechanisms that underlie abuse of alcohol in humans

ELIGIBILITY:
[A] Alcohol use disorders (AUD)

Inclusion Criteria:

1. Males or Females
2. Fulfill DSM5 diagnosis for alcohol use disorder
3. Medically Healthy

Exclusion Criteria:

1. Pregnancy or lactation
2. Comorbid severe/major medical, psychiatric (such as bipolar and psychotic disorders, etc.,) and current comorbid drug use disorders (other than tobacco use and recreational marijuana use)
3. Metal implants or paramagnetic objects contained within the body which may interfere with MRI scans
4. Currently employed as a radiation worker, or participation in radiation drug research procedures within the previous year
5. Currently on any psychotropic medications that can influence nociceptin transmission in the brain

[B]Healthy controls

Inclusion Criteria:

1. Males or females
2. Absence of present or past psychiatric conditions (including alcohol or drug use disorders)
3. Medically Healthy

Exclusion Criteria:

1. Pregnancy of lactation
2. Medical, psychiatric or comorbid drug/alcohol use disorders
3. Metal implants or paramagnetic objects contained within the body which may interfere with the MRI scan
4. Currently employed as a radiation worker; or participation in radioactive drug research protocols within the previous year
5. Currently on any psychotropic medications that can influence nociceptin transmission in the brain
6. Family history of psychotic disorder, manic episode, drug and alcohol use disorder in first-degree relatives

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2016-05-27 (Actual); Primary Completion 2021-03-30 (Actual); Study Completion 2021-03-30 (Actual)

PRIMARY OUTCOMES:
[C-11]NOP-1A VT | Baseline
  VT-Volume of distribution expressed relative to total plasma

CONTACTS AND LOCATIONS:
Locations (1):
- University of PIttsburgh PET Facility, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No